CLINICAL TRIAL: NCT05197218
Title: Prebiotic Properties of Phenolic Compounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR(AG)33/2021
Record Dates: First submitted 2021-11-10; First posted 2022-01-19 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: intestinal gas; healthy subjects; microbiota; prebiotics
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Prebiotic administration
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Combination of a polyphenol rich extract of chokeberry (Aronia melanocarpa) and a polyphenol rich extract of cranberry (Vaccinium macrocarpon Aiton) will be administered for 18 days.

SUMMARY:
Gas evacuated per anus originates by-and-large in the colon, where unabsorbed meal residues are fermented by colonic bacteria. Within subjects, gas output varies in relation to the diet. However, there is a great interindividual variability: gas evacuation in subjects maintained on a similar diet may differ substantially, and this depends on the composition and metabolic pathways of the colonic microbiota. Hence, the volume of gas production and anal evacuation is determined by two main factors: the diet, particularly the amount of fermentable residues, and the individual composition of colonic microbiota. A series of recent studies suggest that some non-absorbable, fermentable meal products (prebiotics) serve as substrate to colonic bacteria and change their composition, thereby producing beneficial effects to the host. These products are fermented by bacteria and at initial intake increase gas production and may induce gas-related symptoms. However, after 7-10 days administration some prebiotics induce an adaptation of intestinal microbiota towards more efficient metabolic pathways with less gas production and the initial symptoms disappear. Some data suggest that phenolic compounds have prebiòtic properties. Aim of the study: to explore the prebiotic effect of a combination of two polyphenol-rich berry extracts (cranberry and chokeberry). Design: single-centre, single arm, open label, proof-of-concept study in healthy subjects. Intervention: a combination of a polyphenol rich extract of chokeberry (Aronia melanocarpa) and a polyphenol rich extract of cranberry (Vaccinium macrocarpon Aiton) will be administered for 18 days. Outcomes: during 2 days immediately before, at the beginning and at the end of the administration phase participants will be put on a standard diet and the following outcomes will be measured: a) number of gas evacuations during daytime for 2 days by means of an event marker; b) perception of digestive sensations by daily scales; c) microbiota composition by fecal analysis; d) metabolites in urine.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* gastrointestinal symptoms
* recent (3 months) antibiotic intake
* change in dietary habits 4 weeks before

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Number of daily anal gas evacuations | 18 days
  Change in the number of anal gas evacuations measured by an event marker from beginning of treatment to end of treatment

SECONDARY OUTCOMES:
Microbiota composition by fecal analysis | 18 days
  Change from beginning of treatment to end of treatment
Sensation of flatulence by scales | 18 days
  Sensation of flatulence measured on a 0-10 scale graded from 0 (no flatulence) to 10 (very intense sensation). Change from beginning of treatment to end of treatment
Sensation of abdominal bloating by scales | 18 days
  Sensation of abdominal bloating measured on a 0-10 scale graded from 0 (no bloating) to 10 (very intense sensation). Change from beginning of treatment to end of treatment.
Sensation of digestive well-being by scales | 18 days
  Sensation of digestive well-being measured on a -5 to +5 scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation). Change from beginning of treatment to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain